CLINICAL TRIAL: NCT06065761
Title: Improving Risk Stratification of Emergency Department Patients With Acute Heart Failure: Building and Testing a Machine-learning Platform for Personalized, Accurate, Real-time Risk Prediction
Brief Title: Improving Risk Stratification of Emergency Department Patients With Acute Heart Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: 1719171
Record Dates: First submitted 2023-09-26; First posted 2023-10-04 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure
Keywords: Emergency Department; Risk Prediction
MeSH Terms: conditions — Heart Failure; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Comprehensive ED heart failure management tool — The investigators plan a regional implementation of an electronic health record-based heart failure decision support tool across 21 EDs of Kaiser Permanente Northern California (KPNC).

SUMMARY:
The primary goal is to build and test a previously developed and validated risk model and clinical decision support tool embedded within the electronic health record to improve risk stratification of emergency department (ED) patients with acute heart failure (AHF).

DETAILED DESCRIPTION:
The study team will build an electronic health record-embedded clinical decision support tool using a recently developed risk prediction model that curates patient-specific data in real-time, accurately estimates short-term patient risk, and presents tailored clinical recommendations. This will be a regional implementation study in which the tool is turned on at 21 emergency departments (ED) across Kaiser Permanente Northern California (KPNC). The study team will validate risk predictions and study key clinical outcomes as part of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18y) KPNC members treated in the ED for presumed acute heart failure

Exclusion Criteria:

* Children (<18y).
* Patients who left against medical advice or eloped prior to ED physician evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to KPNC emergency departments with eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 17459 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with serious adverse events | 30 days from index ED visit
  Serious adverse events include mortality, cardiopulmonary resuscitation (CPR), intubation/ventilation, new end-stage renal disease (ESRD), balloon pump placement, or percutaneous coronary intervention (PCI)/coronary artery bypass grafting (CABG)
Number of patients with all-cause mortality | 30 days from index ED visit

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Kaiser Permanente Antioch Emergency Department, Antioch, California
  - Kaiser Permanente Fremont Emergency Department, Fremont, California
  - Kaiser Permanente Fresno Medical Center, Fresno, California
  - Kaiser Permanente Manteca Medical Center, Manteca, California
  - Kaiser Permanente Modesto Medical Center, Modesto, California
  - Kaiser Permanente Oakland Emergency Department, Oakland, California
  - Kaiser Permanente Redwood City Emergency Department, Redwood City, California
  - Kaiser Permanente Richmond Emergency Department, Richmond, California
  - Kaiser Permanente Roseville Emergency Department, Roseville, California
  - Kaiser Permanente South Sacramento Emergency Department, Sacramento, California
  - Kaiser Permanente Sacramento Emergency Department, Sacramento, California
  - Kaiser Permanente San Francisco Emergency Department, San Francisco, California
  - Kaiser Permanente San Jose Emergency Department, San Jose, California
  - Kaiser Permanente San Leandro Emergency Department, San Leandro, California
  - Kaiser Permanente San Rafael Emergency Department, San Rafael, California
  - Kaiser Permanente Santa Clara Emergency Department, Santa Clara, California
  - Kaiser Permanente Santa Rosa Emergency Department, Santa Rosa, California
  - Kaiser Permanente South San Francisco Emergency Department, South San Francisco, California
  - Kaiser Permanente Vacaville Medical Center, Vacaville, California
  - Kaiser Permanente Vallejo Medical Center, Vallejo, California
  - Kaiser Permanente Walnut Creek Medical Center, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: No